CLINICAL TRIAL: NCT00340652
Title: Study of Estrogen Activity & Development (SEAD) - SEAD 1 Sonography
Brief Title: Effects of Infant Diets on Estrogen Activity and Development
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903287; 03-E-N287
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2012-08-22

CONDITIONS: Hormone
Keywords: Soy; Isoflavones; Infant Formula; Sexual Development; Hormone

SUMMARY:
This study, conducted at the Children's Hospital of Boston and the Brigham and Women's Hospital in Boston, will examine the natural history of infant development in the first year of life and how different types of infant feeding may affect that development. During pregnancy, babies are exposed to the female hormone estrogen from their mothers. Estrogen affects development of breasts and milk production, as well as the development of the uterus, ovaries and possibly other hormonally responsive organs in both males and females. Between 6 and 12 months of age, the effects are reduced. Breast milk and some infant formulas may contain compounds that can act like female hormones in the body and may prolong the estrogen effects. This study will examine the natural history of estrogen activity in infants on different feeding regimens, breast milk, cow's milk, and soy milk and will serve as preparation for a larger study of the effects of soy formula on estrogen activity in infants.

Full-term female babies (37 to 41 weeks gestational age at birth) from 0 to 12 months of age and male babies from birth to 6 months of age who weigh from 2501 to 4499 grams (about 5.5 to 10 pounds) at birth and who have no chromosomal abnormalities, major malformations, or endocrine problems may be eligible for this study. Males must have palpable testes. Babies being fed a diet of breast milk, soy milk, or cow's milk will be included. Study procedures include the following:

* History of the baby's dietary intake since birth, provided by the parent;
* Ultrasound measurement of the uterus, ovaries, and breasts in female babies; the testes, prostate, and breasts in males; and the thymus, thyroid, and kidneys in all babies;
* Measurements of all babies' weight, length, and head circumference.

DETAILED DESCRIPTION:
Term newborns have anatomic and sonographic evidence of in utero estrogen exposure. Over the first six months to a year of life, as the influence of maternal hormone wanes, these findings recede. Soy infant formula contains large amounts of isoflavones (daidzein and genistein) that can occupy estrogen receptors and act as estrogens in the laboratory. A food substance with estrogen activity might prolong the effect of maternal hormones, or interfere with hormonal homeostasis in the child. This cross-sectional pilot study will be undertaken in order to establish methods for a future multi center study designed to assess the potential effects of soy formula on estrogen activity in infants. In this pilot study (SEAD 1), 156 examinations on full-term infants, ages 0-12 months and on one of three feeding regimens (soy formula, breast milk or cow's milk formula) will be completed to see if their exposure to soy estrogen compared to breast milk and non-soy formulas prolongs anatomical evidence of estrogen exposure and response. A schedule of visits for SEAD 1 is included in Appendix A. In addition to SEAD 1, two other cross-sectional studies (SEAD 2 and SEAD 3) will be undertaken to evaluate anatomical evidence by physical examination (SEAD 2) and assess the hormonal and biochemical status of full-term infants ages 0-12 months (SEAD 3). These studies will be conducted at Children's Hospital of Philadelphia (CHOP) in parallel with the SEAD 1 study. Further details of SEAD 2 and 3 will not be presented in this protocol. The purpose of the SEAD 1 pilot study is twofold. The first is to develop and finalize recruitment and collections procedures in preparation for a larger, comprehensive trial of biological response in children to soy formula with and without the estrogenic isoflavones. The second is to study the natural history of estrogen activity in infants on a variety of feeding regimens.

ELIGIBILITY:
* INCLUSION CRITERIA:

Full term infants defined as age 37-41 weeks gestational age at birth. Ultrasound evidence or reliable reporting of last menstrual period (LMP) by infant's mother.

Can be categorized into one of the feeding definitions:

Breastmilk Category:

0-48 hours old (Age-Interval: 1) - Breastmilk exclusively;

49 hours - 3 months (Age-Interval: SEAD1 = 2 through 7) - Breastmilk exclusively;

Greater than 3 months (Age-Interval: SEAD1 = 8 through 19) - Breastmilk exclusively OR Breastmilk and Cow-based formula.

Restriction: Babies in the Breastmilk category are not allowed to have had any SOY foods including SOY formula and solid foods containing SOY in their lifetime.

Cow-Based Formula Category:

0-48 hours old (Age-Interval: 1) - Cow-based formula exclusively;

49 hours - 3 months (Age-Interval: SEAD1 = 2 through 7) - Cow-based formula exclusively;

Greater than 3 months (Age-Interval: SEAD1 = 8 through 19) - Cow-based formula exclusively.

Exception: If a baby was Breastfed in the nursery, the baby must have gone home on Cow-based formula and have been on Cow-based formula exclusively ever since. Such a child cannot participate in the SEAD study until s/he has been exclusively Cow-based formula fed for at last 2 weeks.

Restriction: Babies in the Cow-based formula category are not allowed to have had any SOY foods including SOY formula and solid foods containing SOY in their lifetime.

Soy Formula Category:

0-48 hours old (Age-Interval: 1) - Soy formula exclusively;

49 hours - 3 months (Age-Interval: SEAD1 = 2 through 7) - Soy formula exclusively;

Greater than 3 months (Age-Interval: SEAD1 = 8 through 19) - 2/3 of lifetime on Soy formula exclusively & continuously, and including the two weeks up to the exam.

Exception: If a baby was fed something other than Soy formula in the nursery, the baby must have gone home on Soy and been on Soy exclusively ever since. Such a child cannot participate in the SEAD study until s/he has been exclusively Soy-fed for at least 2 weeks.

Birth weight between 2501 - 4499 grams.

Age 0-12 months for girls and age 0-6 months for boys.

EXCLUSION CRITERIA:

Chromosomal anomalies.

Major malformations.

Non-palpable testis (males only).

Presence of an endocrinopathy (i.e., ambiguous genitalia, congenital hypothyroidism).

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 157 (Actual)
Dates: Start 2003-08-26; Study Completion 2012-08-22

CONTACTS AND LOCATIONS:
Overall Officials: Walter Rogan, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Childrens Hospital, Boston, Boston, Massachusetts

REFERENCES:
- [Background] Setchell KD, Zimmer-Nechemias L, Cai J, Heubi JE. Isoflavone content of infant formulas and the metabolic fate of these phytoestrogens in early life. Am J Clin Nutr. 1998 Dec;68(6 Suppl):1453S-1461S. doi: 10.1093/ajcn/68.6.1453S. PMID 9848516
- [Background] Cruz ML, Wong WW, Mimouni F, Hachey DL, Setchell KD, Klein PD, Tsang RC. Effects of infant nutrition on cholesterol synthesis rates. Pediatr Res. 1994 Feb;35(2):135-40. doi: 10.1203/00006450-199402000-00001. PMID 8165045
- [Background] Strom BL, Schinnar R, Ziegler EE, Barnhart KT, Sammel MD, Macones GA, Stallings VA, Drulis JM, Nelson SE, Hanson SA. Exposure to soy-based formula in infancy and endocrinological and reproductive outcomes in young adulthood. JAMA. 2001 Aug 15;286(7):807-14. doi: 10.1001/jama.286.7.807. PMID 11497534